CLINICAL TRIAL: NCT06421883
Title: The Potential Impact of Probiotic Supplementation on Trimethylamine-N-Oxide Plasma Level in End Stage Renal Disease Patients Undergoing Hemodialysis
Brief Title: Study the Effect of Probiotic Supplementation on Trimethylamine-N-Oxide Plasma Level in Hemodialysis Patients
Acronym: probiotic
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Nehal Kamal Bazid, Principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Interventional clinical trial
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: End Stage Renal Disease
Keywords: hemodialysis; probiotic; Trimethylamine-N-Oxide; TMAO
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups each group includes 40 patients:
  Control group: 40 patients will receive their standard therapy only. Intervention group (probiotic group): 40 patients will receive probiotic 5 billion unit per day with their standard therapy for 3 months.
Masking Description: (Open Label)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental probiotic group (Experimental): Experimental probiotic group patients will receive probiotic 5 billion unit per day with their standard therapy collect blood sample and measure TMAO at baseline and after 3 months
  Interventions: Dietary Supplement: Lactobacillus containing probiotic
- control group (No Intervention): No Intervention: control group patients will receive their standard therapy only collect blood sample and measure TMAO at baseline and after 3 months

INTERVENTIONS:
Dietary Supplement: Lactobacillus containing probiotic — Patients will be randomized into two groups each group includes 40 patients:
  Control group: 40 patients will receive their standard therapy only. Intervention group (probiotic group): 40 patients will receive probiotic 5 billion unit per day with their standard therapy for 3 months.
  Other Names: probiotic
  Arms: Experimental probiotic group

SUMMARY:
The goal of this clinical trial is to learn if probiotic has an effect on Trimethylamine-N-Oxide Plasma Level in plasma, which represent strong risk factor for Atherosclerosis in end stage renal disease patients who undergoing hemodialysis the main questions to answer are : Does probiotic lower Trimethylamine-N-Oxide concentration? does probiotic participating in decreasing risk of atherosclerosis in end stage renal disease patients undergoing hemodialysis ? research will compare between patients who are taking probiotic and control group (taking no drug) participants will take probiotic for 3 months visit the clinic once every 2 weeks for checkups and tests

All Patients will be subjected to the following:

1. Informed consent.
2. Demographics and history taking: Using Patient Data sheet.
3. Laboratory evaluation including:

Kidney function tests: blood urea,serum creatinine, albumin ,uric acid. Complete blood count (CBC).

C-reactive protein (CRP).

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD) is considered as a major public health problem as it can lead to end-stage kidney failure, which requires replacement therapy. A prompt and accurate diagnosis, along with the appropriate treatment, can delay CKD's progression End-stage renal disease (ESRD) is associated with significant alterations in cardiovascular function; homeostasis of body fluid, electrolytes, and acid-base equilibrium; bone metabolism, erythropoiesis; and blood coagulation. The prevalence of ESRD is increasing rapidly worldwide, as is the number of patients requiring surgery under general anesthesia. Patients with ESRD have significantly higher risks of perioperative morbidity and mortality due to multiple comorbidities Trimethylamine N-oxide (TMAO) is a gut microbiota metabolite derived from trimethylamine containing nutrient precursors such as choline, L-carnitine, and betaine. An increasing number of clinical studies have demonstrated a strong relationship between elevated plasma TMAO levels and adverse cardiovascular events. It is commonly agreed that TMAO acts as both an independent risk factor and a prognostic index for patients with cardiovascular disease , TMAO is considered as a potential biomarker and/or therapeutic target for diagnosis and treatment of patients with cardiovascular disease Probiotic work as antagonist for those strains which are responsible for the synthesis of TMAO precursor molecules in the gut and modulate miRNAs associated with the genes which are responsible for TMA lyases and ultimately play a role in conversion of diet precursor into TMA Control group: 40 patients will receive their standard therapy only. Intervention group (probiotic group): 40 patients will receive probiotic 5 billion unit per day with their standard therapy for 3 months

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed as End Stage Renal Disease with hemodialysis
* Aged 18 years or older.
* Both sexes.
* No known contraindications to therapy with probiotic
* Patients who accept to participate in the study.

Exclusion Criteria:

* Pregnant and breast-feeding women
* History of severe allergic reactions to the study medication.
* Current medication regimen including probiotic
* chronic liver disease
* Patients receiving chronic anti-inflammatory therapy
* Non-compliant patients: those who did not adhere to the medications during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
change in Trimethylamine-N-Oxide Plasma Level | 3 months
  probiotic is expected to lower Trimethylamine-N-Oxide Plasma Level in dialysis patients

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No